CLINICAL TRIAL: NCT07205926
Title: First-in-human, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study Evaluating the Safety and Immunogenicity of IVT Shigella-04 in Healthy Young Adults
Brief Title: First in Human Dose Escalation Study Evaluating the Safety and Immunogenicity of IVT's Shigella-04 Vaccine in Healthy Young Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inventprise Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IVT 514
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Shigella; Diarrhea
MeSH Terms: conditions — Dysentery, Bacillary; Diarrhea | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects are randomized in five groups in a 5:1, each receiving 2-doses of IVT Shigella-04 or placebo.
Who Masked: Participant, Investigator
Masking Description: Subjects and investigators will be blinded to treatment assignment. The vaccine and placebo will be prepared and administered by dedicated unblinded staff not involved in other aspects of the study and will be concealed from the participant at the time of dosing. Unblinding will occur only after database lock or in the event of a medical emergency requiring knowledge of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Shigella-04 Low Dose without adjuvant (0.5 mL dose) (Experimental): Subjects will receive a 0.5 mL dose of the Shigella-04 low-dose formulation of each conjugated OPS, and administered via intramuscular injection on Day 1 and 29
  Interventions: Biological: IVT Shigella-04
- Shigella-04 Low Dose with adjuvant (0.5 mL dose) (Experimental): Subjects will receive a 0.5 mL dose of the Shigella-04 low-dose formulation of each conjugated OPS, with adjuvant, administered via intramuscular injection on Day 1 and 29
  Interventions: Biological: IVT Shigella-04
- Shigella-04 Medium Dose without adjuvant (0.5 mL dose) (Experimental): Subjects will receive a 0.5 mL dose of the Shigella-04 medium-dose formulation of each conjugated OPS, and administered via intramuscular injection on Day 1 and 29
  Interventions: Biological: IVT Shigella-04
- Shigella-04 Medium Dose with adjuvant (0.5 mL dose) (Experimental): Subjects will receive a 0.5 mL dose of the Shigella-04 medium-dose formulation of each conjugated OPS, with adjuvant, administered via intramuscular injection on Day 1 and 29
  Interventions: Biological: IVT Shigella-04
- Shigella-04 High Dose without adjuvant (1.0 mL dose) (Experimental): Subjects will receive a 1.0 mL dose of the Shigella-04 high-dose formulation of each conjugated OPS, and administered via intramuscular injection on Day 1 and 29
  Interventions: Biological: IVT Shigella-04
- Placebo - 0.9% Saline (Placebo Comparator): 0.9% saline
  Interventions: Biological: Placebo (0.9% saline)

INTERVENTIONS:
Biological: IVT Shigella-04 — Preventative vaccine for Shigella protection against 4 unique serotypes
  Arms: Shigella-04 High Dose without adjuvant (1.0 mL dose); Shigella-04 Low Dose with adjuvant (0.5 mL dose); Shigella-04 Low Dose without adjuvant (0.5 mL dose); Shigella-04 Medium Dose with adjuvant (0.5 mL dose); Shigella-04 Medium Dose without adjuvant (0.5 mL dose)
Biological: Placebo (0.9% saline) — Subjects dosed with 0.9% saline
  Other Names: Placebo
  Arms: Placebo - 0.9% Saline

SUMMARY:
Phase 1 trial to evaluate the Safety and Immunogenicity of Inventprise's (IVT) Shigella-04 in Healthy Young Adults

DETAILED DESCRIPTION:
A phase 1 single-site, randomized, double-blind, placebo-controlled, dose-escalation clinical trial to evaluate the safety and immunogenicity of a 2-dose regimen of IM injection of 5 dose formulations of IVT Shigella-04 vaccine with and without adjuvant among 60 healthy individuals aged 18 to 49 years. Approximately 12 eligible participants will be enrolled in the specified 5 sequential dose cohorts and randomized in a 5:1 ratio to receive 2 IM injections of IVT Shigella-04 or placebo (normal saline) at a 28-day interval.

ELIGIBILITY:
Inclusion Criteria

Participants who meet all the following criteria may be included in the study:

1. Age 18 to 49 years at the time of Dose 1
2. Good general health status, as determined by medical history, physical examination, safety laboratory tests, ECG, vital signs, and clinical judgment
3. BMI ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2
4. Negative alcohol breath test and urine drug screen results at Screening and on Day 1
5. All women: negative serum pregnancy test at Screening and negative urine pregnancy on Day 1
6. Women of childbearing potential (see definition in Section 6.6.1): willingness to use a highly effective form of contraception (see list in Section 6.6.1) through 28 days after the last IP dose
7. Willingness to attend all protocol visits and to have all protocol-required procedures
8. Provision of written informed consent

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from the study:

1. Currently lactating
2. History of shigellosis or participation in a Shigella challenge study
3. History of bloody diarrhea without alternative diagnosis
4. History of inflammatory bowel disease
5. History of anaphylaxis or angioedema
6. History of malignancy, excluding nonmelanoma skin cancer, cervical carcinoma in situ, and malignancies considered cured > 5 years prior to Day 1
7. History of diabetes mellitus (Individuals with diet-controlled diabetes or history of gestational diabetes are eligible if screening blood glucose is normal and there has been no requirement for antidiabetic medication in the last year.)
8. Known hypersensitivity to any of the ingredients in IVT Shigella-04
9. Inadequate venous access for repeated phlebotomy
10. Any screening laboratory test result outside the normal range and grade ≥ 2 according to the FDA's toxicity grading scale for vaccine trials in healthy adults and adolescents; (Elevated creatine kinase and isolated elevations of bilirubin may be Grade 2 if hepatic transaminases are normal and the Investigator attributes the abnormality to exercise or Gilbert's syndrome. Potential cases of benign ethnic neutropenia should be discussed with the Medical Monitor)
11. Positive serologic test for human HIV-1 or HIV-2 antibody, hepatitis B surface antigen, or hepatitis C antibody
12. Immunodeficiency or chronic administration (> 14 consecutive days) of immunosuppressant or other immune-modifying drugs (see details in Section 6.6.2), including systemic glucocorticoids, within 6 months before Day 1 (topical, intra-articular, or inhaled glucocorticoids permitted)
13. Previous receipt of a licensed or investigational Shigella vaccine
14. Planned receipt of any other vaccine through Day 57
15. Receipt of blood transfusion or blood product within 6 months before Day 1 or planned receipt through Day 57
16. Receipt of any other IP within 90 days before Day 1 or planned receipt through the end of the study
17. Planned elective hospitalization or surgical procedure through the end of the study
18. Occupational exposure to Shigella (eg, laboratory work)
19. Residence ≥ 6 months in a low-income or lower-middle-income country as defined by the World Bank (https://datatopics.worldbank.org/world-development-indicators/the-world-by-income-and-region.html)
20. Employee of Inventprise, vendors, or research sites associated with the study
21. Any medical, psychiatric, substance use, or social condition that, in the judgment of the Investigator, may pose a risk to the participant or interfere with protocol adherence, assessment of study objectives, or ability to provide informed consent

Temporary Delay Criteria

Administration of IVT Shigella-04/placebo will be delayed for any participant who meets any of the following criteria:

1. Receipt of any vaccine in the past 7 days
2. Febrile illness (eg, oral temperature ≥ 38.0°C), diarrhea, or other acute illness in the past 48 hours
3. Presence of any other sign, symptom, or medication use that could inhibit the proper vaccine administration of IVT Shigella-04/placebo or interpretation of diary data

These criteria are temporary or self-limiting, and IVT Shigella-04/placebo may be administered once the time frame has elapsed/the condition has resolved.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with reactogenicity events for 7 days after each dose | 7 days after Doses 1 and 2
  To assess the safety and tolerability of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Percentage of participants with adverse events (AEs) from Dose 1 to 28 days after Dose 2 | After Dose 1 to 6 months after Dose 2
  To assess the safety and tolerability of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Percentage of participants with medically attended AE's (MAAEs) from Dose 1 to 6 months after Dose 2 | After Dose 1 to 6 months after Dose 2
  To assess the safety and tolerability of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Percentage of participants with newly diagnosed chronic medical conditions (NDCMCs) from Dose 1 to 6 months after Dose 2 | After Dose 1 to 6 months after Dose 2
  To assess the safety and tolerability of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Percentage of participants with AEs of special interest (AESIs) from Dose 1 to 6 months after Dose 2 | After Dose 1 to 6 months after Dose 2
  To assess the safety and tolerability of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Percentage of participants with serious AEs (SAEs) from Dose 1 to 6 months after Dose 2 | After Dose 1 to 6 months after Dose 2
  To assess the safety and tolerability of a 2-dose IM regimen of 5 formulations of IVT Shigella-04

SECONDARY OUTCOMES:
Percentage of participants achieving 4-fold increase in anti-IpaB and serotype-specific anti-OPS immunoglobulin G (IgG) concentration at 28 days after each dose and 6 months after Dose 2 | At 28 days after each dose and 6 months after Dose 2
  To assess the humoral immunogenicity of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Geometric mean concentration (GMCs) of anti-IpaB and serotype-specific anti-OPS IgG at 28 days after each dose and 6 months after Dose 2 | At 28 days after each dose and 6 months after Dose 2
  To assess the humoral immunogenicity of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Geometric mean fold rises (GMFRs) in anti-IpaB and serotype-specific anti-OPS IgG concentration at 28 days after each dose and 6 months after Dose 2 | At 28 days after each dose and 6 months after Dose 2
  To assess the humoral immunogenicity of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Percentage of participants achieving 4-fold increase in serotype-specific anti-OPS functional antibody titer measured by serum bactericidal assay (SBA) at 28 days after each dose | At 28 days after each dose
  To assess the humoral immunogenicity of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
Geometric mean titers (GMTs) of serotype-specific anti-OPS functional antibody as measured by SBA at 28 days after each dose | At 28 days after each dose
  To assess the humoral immunogenicity of a 2-dose IM regimen of 5 formulations of IVT Shigella-04
GMFRs in serotype-specific anti-OPS functional antibody titer as measured by SBA at 28 days after each dose | At 28 days after each dose
  To assess the humoral immunogenicity of a 2-dose IM regimen of 5 formulations of IVT Shigella-04

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Inventprise Inc.
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code